CLINICAL TRIAL: NCT07111611
Title: Effects of Non-Traumatic Nasopharyngeal Suction Technique in Infants During Non-Invasive Ventilation
Brief Title: Effects of Non-Traumatic Nasopharyngeal Suction Technique in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, ebru temizsoy, Phd, Istanbul Bilgi University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 159
Record Dates: First submitted 2025-05-25; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Preterm
Keywords: non-invasive ventilation; preterm infant; suction; pain; physological parameters
MeSH Terms: conditions — Premature Birth; Pain

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Randomized Controlled two groups (control group and study group)
Who Masked: Investigator
Masking Description: Single (Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Traumatic Suction Group (Experimental): Infants in this group underwent a non-traumatic oro/nasopharyngeal suction procedure. A 10 Fr suction catheter with a blunt-cut tip and a 10 ml syringe were used. Depending on secretion amount and thickness, 5-10 ml of 0.9% saline was rapidly instilled through one nostril. Secretions were then aspirated using 150-200 mmHg negative pressure via the opposite nostril and the mouth, without deep catheter insertion.
  Physiological parameters (heart rate, respiratory rate, oxygen saturation, skin color) and behavioral responses (N-PASS pain and sedation scores) were recorded before, during, and 10 minutes after the procedure.opposite nostril and the mouth, without deep catheter insertion. The procedure was carefully performed without mucosal contact to prevent trauma and bleeding. The entire aspiration process lasted 5-10 seconds. Physiological parameters and behavioral responses (N-PASS scores) were recorded before, during, and 10 minutes after the procedure.
  Interventions: Procedure: Non-Traumatic Nasopharyngeal Suction Procedure
- Standard Suction Group (No Intervention): Infants in this group received routine oro/nasopharyngeal suctioning as performed in standard clinical practice.
  A 6-8 Fr suction catheter was used without prior saline instillation. The catheter was inserted through the mouth and/or nostrils into the nasopharynx, and secretions were aspirated using 60-100 mmHg negative pressure.
  The suction procedure lasted 5-10 seconds. The same physiological and behavioral parameters were monitored and recorded before, during, and after the procedure.

INTERVENTIONS:
Procedure: Non-Traumatic Nasopharyngeal Suction Procedure — A modified suctioning technique that avoids deep catheter insertion and minimizes mucosal contact. Sterile saline (0.9%) is instilled into one nostril, and secretions are aspirated using external suction via the opposite nostril or mouth. This approach is designed to reduce pain and physiological stress compared to standard suction methods in preterm infants undergoing non-invasive ventilation.
  Other Names: Non-traumatic Suction Technique
  Arms: Non-Traumatic Suction Group

SUMMARY:
Background: Non-invasive ventilation (NIV) in preterm infants often leads to secretion-related airway obstructions, requiring suctioning. Traditional oro/nasopharyngeal suction techniques may cause mucosal trauma, pain, and physiological instability.

Objective: To evaluate the effects of a novel non-traumatic oro/nasopharyngeal suction technique on physiological and behavioral parameters in preterm infants receiving NIV.

Methods: A randomized controlled trial was conducted with 100 preterm infants (32 0/6 - 36 6/7 weeks gestation) admitted to a Level IV NICU. Infants were randomized into intervention (non-traumatic suction) and control (routine suction) groups. Data on heart rate, respiratory rate, SpO₂, skin color, and pain/sedation scores (N-PASS) were collected before, during, and after suctioning.

DETAILED DESCRIPTION:
This randomized controlled clinical trial was conducted to evaluate the effectiveness of a newly developed non-traumatic oro/nasopharyngeal suction technique in preterm infants receiving non-invasive ventilation (NIV). Traditional suction methods used to remove airway secretions in neonates are often associated with complications such as mucosal trauma, bradycardia, hypoxia, and increased pain.

The non-traumatic technique involves administering a small volume of sterile saline through one nostril and using gentle suction from the other nostril or the mouth without direct mucosal contact. This approach is designed to minimize trauma and discomfort.

A total of 100 preterm infants with gestational ages between 32 0/6 and 36 6/7 weeks were included and randomized into two groups: an intervention group receiving the non-traumatic suction method and a control group undergoing standard suction. Key outcome measures included physiological parameters (heart rate, respiratory rate, SpO₂, skin color) and behavioral indicators assessed using the Neonatal Pain, Agitation, and Sedation Scale (N-PASS). Data were collected before, during, and after suctioning procedures.

ELIGIBILITY:
Inclusion Criteria:

Gestational age between 32 0/6 and 36 6/7 weeks

Receiving non-invasive ventilation (NIV) via nasal CPAP

Clinically stable prior to suctioning

Parental or legal guardian informed consent obtained

Age within first 7 days of life at time of first suction procedure

Exclusion Criteria:

Major congenital anomalies (e.g., craniofacial malformations, cardiac defects)

Suspected or confirmed neurological disorders (e.g., intraventricular hemorrhage Grade III/IV)

Presence of upper airway obstruction or nasal anomalies

Infants requiring invasive mechanical ventilation at the time of study

Any condition requiring continuous sedation or analgesia

Hemodynamically unstable infants (e.g., hypotension requiring inotropes)

Parental refusal or withdrawal of consent

Ages: 32 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Change in Pain Score During Suctioning, N-PASS (Neonatal Pain, Agitation, and Sedation Scale) pain subscore | During suctioning (within 1 minute of procedure start)
  To evaluate and compare the level of pain experienced by preterm infants during suctioning using either the non-traumatic or standard technique. Pain Subscore: Range = 0 to 10, higher score = more pain.

SECONDARY OUTCOMES:
Change in Oxygen Saturation (SpO₂) During and After Suctioning | During suctioning and 10 minutes post-procedure. SpO₂ measured by pulse oximetry.
  To assess the impact of suction technique on oxygenation stability.
Change in Heart Rate (HR) During and After Suctioning | During suctioning and 10 minutes post-procedure. Heart Rate measured using bedside monitor.
  To compare the effect of suction methods on cardiovascular stability.
Change in Sedation Score During Suctioning,N-PASS sedation subscore, | During suctioning
  To measure the behavioral reponse and comfort level of the infant during the procedure. Sedation Subscore: Range = -2 to +2, lower = deeper sedation

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Temizsoy, PhD,RN, Principal Investigator — İstanbul Bilgi University
Locations (1):
- İstanbul Bilgi University, Şişli, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No